CLINICAL TRIAL: NCT06190951
Title: A Phase 2 Peri-operative Trial of Fianlimab and Cemiplimab Compared With Anti-PD1 Alone in Patients With Resectable Stage III and IV Melanoma
Brief Title: A Trial to Learn if Fianlimab and Cemiplimab Are Safe and Work Better Than Anti-PD1 Alone in Adult Participants With Resectable Stage 3 or 4 Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R3767-ONC-2208; 2022-502825-17-00 (EU CTIS Number)
Record Dates: First submitted 2023-11-09; First posted 2024-01-05 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Melanoma
Keywords: Skin cancer; Fully resectable stage III melanoma; Fully resectable stage IV melanoma
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — cemiplimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (Active Comparator): As described in the protocol
  Interventions: Drug: cemiplimab; Drug: Placebo
- Arm B (Experimental): As described in the protocol
  Interventions: Drug: Fixed Dose Combination (FDC) cemiplimab+fianlimab
- Arm C (Experimental): As described in the protocol
  Interventions: Drug: Fixed Dose Combination (FDC) cemiplimab+fianlimab

INTERVENTIONS:
Drug: cemiplimab — Administered per the protocol
  Other Names: REGN2810; Libtayo
  Arms: Arm A
Drug: Fixed Dose Combination (FDC) cemiplimab+fianlimab — Or coadministration, depending on availability.
  Other Names: REGN2810; Libtayo; REGN3767
  Arms: Arm B; Arm C
Drug: Placebo — Administered per the protocol
  Arms: Arm A

SUMMARY:
This study is researching an experimental drug called REGN3767, also known as fianlimab (R3767), when combined with another medication called cemiplimab (each individually called a "study drug" or called "study drugs" when combined) compared with cemiplimab alone. These types of immunotherapy study drugs are collectively known as immune checkpoint inhibitors. Immunotherapies are treatments that use the immune system to recognize and kill cancer cells. The study is focused on participants with a type of skin cancer known as melanoma.

The objective of this study is to see if the combination of fianlimab and cemiplimab is an effective treatment compared to cemiplimab in participants with high-risk, resectable melanoma. Participants will receive treatment before surgery, undergo resection, and then will have the option to continue treatment after resection.

The study is looking at several other research questions, including:

* What side effects may happen from receiving the study drug(s).
* How much study drug(s) is in the blood at different times.
* Whether the body makes antibodies against the study drug(s) (which could make the drug less effective or could lead to side effects). Antibodies are proteins that are naturally found in the blood stream that fight infections.
* How administering the study drugs might improve quality of life.

ELIGIBILITY:
Key Inclusion Criteria:

1. All patients must be either stage III (IIIB, IIIC, IIID) or stage IV (M1a, M1b, M1c) per American Joint Committee on Cancer (AJCC) 8th edition (Amin 2017) and have histologically confirmed cutaneous melanoma that is deemed completely surgically resectable in order to be eligible as described in the protocol.
2. Patients with stage III melanoma must have clinically detectable disease that is confirmed as malignant on the pathology report. The pathology report must be reviewed, signed and dated by the investigator; this process will be confirmed during the interactive voice response system (IVRS) process as described in the protocol.
3. Patients must be candidates for full resection with curative intent and must be able to be surgically rendered free of disease with negative margins on resected specimens at surgery. The treatment plan including date of surgery must be documented by the investigator prior to randomization.
4. All patients must undergo full disease staging through a complete physical examination and imaging studies within 4 weeks prior to randomization. Imaging must include a computer tomography (CT) scan of the chest, abdomen, pelvis (if the primary tumor is on the head/neck then include a CT scan of head/neck), and all known sites of previously resected disease (if applicable) and brain magnetic resonance imaging (MRI) (or brain CT with contrast allowed if MRI is contraindicated).
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1

Key Exclusion Criteria:

Medical conditions:

1. Primary uveal melanoma
2. Ongoing or recent (within 2 years) evidence of an autoimmune disease that required systemic treatment with immunosuppressive agents. The following are non-exclusionary: vitiligo, childhood asthma that has resolved, residual hypothyroidism that requires only hormone replacement, psoriasis not requiring systemic treatment.
3. Patients must not have received any prior systemic anti-cancer therapy for melanoma. Prior radiotherapy for melanoma is allowed if not given to a target lesion or, if given to a target lesion, there is pathological evidence of disease progression in the same lesion.
4. Uncontrolled infection with human immunodeficiency virus (HIV), hepatitis B (HBV) or hepatitis C virus (HCV) infection; or diagnosis of immunodeficiency that is related to or results in chronic infection as described in the protocol.

   Prior/concomitant therapy:
5. Use of immunosuppressive doses of corticosteroids (≥10mg of prednisone per day or equivalent) within 14 days of the first dose of study medication as described in the protocol.
6. Treatment with any anti-cancer therapy for malignancies other than melanoma, including immuno- therapy, chemotherapy, radiotherapy, or biological therapy in the 5 years prior to randomization as described in the protocol.

   Other comorbidities:
7. Participants with a history of myocarditis.
8. History or current evidence of significant (CTCAE grade ≥2) local or systemic infection (e. g., cellulitis, pneumonia, septicemia) requiring systemic antibiotic treatment within 2 weeks prior to the first dose of trial medication.

Note: Other protocol-defined inclusion/ exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2024-09-18 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2030-12-09 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate as assessed by Blinded Independent Pathological Review (BIPR) | Up to 1 year

SECONDARY OUTCOMES:
pCR rate as assessed by local pathologic review | Up to 1 year
Event-Free Survival (EFS) | Up to 4 years
Distant metastasis-free survival (DMFS) | Up to 4 years
Overall survival (OS) | Up to 4 years
Major pathological response (MPR) as assessed by BIPR | Up to 4 years
MPR rate as assessed by local pathologic review | Up to 4 years
Objective Response Rate (ORR) assessed by investigator per RECIST 1.1 criteria | Up to 4 years
ORR assessed by Blinded Independent Central Review (BICR) per RECIST 1.1 criteria | Up to 4 years
Relapse-free survival (RFS) | Up to 4 years
Occurrence of treatment-emergent adverse events (TEAEs) | 90 days following last dose of study drug, approximately 4 years
Occurrence of immune-mediated adverse events (imAEs) | 90 days following last dose of study drug, approximately 4 years
Occurrence of serious adverse events (SAEs) | 90 days following last dose of study drug, approximately 4 years
Occurrence of adverse events of special interest (AESIs) | 90 days following last dose of study drug, approximately 4 years
Occurrence of TEAEs resulting in death | 90 days following last dose of study drug, approximately 4 years
Occurrence of interruption or discontinuation of study drug(s) due to TEAE. | 90 days following last dose of study drug, approximately 4 years
Occurrence of cancellation of surgery due to TEAE or delay to surgery | 90 days following last dose of study drug, approximately 4 years
Occurrence of laboratory abnormalities | 90 days following last dose of study drug, approximately 4 years
  Grade 3 or higher per Common Terminology Criteria for Adverse Events (CTCAE V5.0)
Concentrations of fianlimab in serum | Up to 4 years
Concentrations of cemiplimab in serum | Up to 4 years
Anti-drug antibodies (ADA) in serum to fianlimab | Up to 4 years
ADA in serum to cemiplimab | Up to 4 years
Change from baseline in disease-related symptoms per Functional Assessment of Cancer Therapy-Melanoma (FACT-M) subscale | Up to 4 years
  The FACT-M is a melanoma-specific quality of life questionnaire that is composed of items from the Functional Assessment of Cancer Therapy-General (FACT-G). The FACT-M is scored on a 5-point Likert-scale: "Not at all", "A little bit", "Somewhat", "Quite a bit", and "Very much.". A Higher score represents higher Health Related Quality of Life (HRQoL).
Change from baseline in functioning per European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (QoL) C30 (EORTC QLQ-C30) | Up to 4 years
  EORTC-QLQ-C30 is a 30-item subject self-report questionnaire composed of both multi-item and single scales, including a global health status/quality of life (GHS/QoL) scale. Participants rate items on a four-point scale, with 1 as "not at all" and 4 as "very much." A change of 5 - 10 points is considered a small change. A change of 10 - 20 points is considered a moderate change.
Change from baseline in global health status/QoL per EORTC QLQ-C30 | Up to 4 years
Change from baseline in overall health state per European Quality of Life Dimension 5 (EQ-5D-5L) | Up to 4 years
  The EQ-5D-5L consists of EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (104):
- United States (28):
  - UC San Diego, La Jolla, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Family Cancer Institute, Newport Beach, California
  - California Pacific Medical Center Research Institute, San Francisco, California
  - University of California San Francisco (UCSF), San Francisco, California
  - St John's Cancer Institute, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Yale University Cancer Center, New Haven, Connecticut
  - Emory Healthcare, Emory Clinic, Atlanta, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute Brookline Avenue, Boston, Massachusetts
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Northwell Health Cancer Institute, Lake Success, New York
  - Duke Cancer Institute, University Hospital, Durham, North Carolina
  - Seidman Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University James Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - UT Southwestern/Simmons Comprehensive Cancer Center, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
- Australia (11):
  - Lismore Base Hospital, Lismore, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Melanoma Institute of Australia, Wollstonecraft, New South Wales
  - The Townsville Hospital, Douglas, Queensland
  - Hervey Bay Hospital, Hervey Bay, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Icon Cancer Centre Hobart, Hobart, Tasmania
  - Eastern Health, Box Hill, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - One Clinical Research at Hollywood Private Hospital, Nedlands, Western Australia
- Austria (4):
  - University Hospital Saint Poelten, Sankt Pölten, Lower Austria
  - Medical University of Graz, Graz, Styria
  - Medical University Innsbruck, Innsbruck, Tyrol
  - Medical University of Vienna, Vienna
- Canada (4):
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal (CHUM), Montreal, Quebec
  - CHU de Quebec - Universite Laval, Québec
- France (16):
  - Hospices Civils de Lyon, Pierre-Bénite, Auvergne-Rhône-Alpes
  - Centre Georges Francois Leclerc, Dijon, Bourgogne-Franche-Comté
  - CHU-Dijon, Dijon, Burgundy
  - CHRU de Tours, Tours, Centre-Val de Loire
  - Chu De Bordeaux, Bordeaux, Gironde
  - Centre Hospitalier Universitaire Grenoble Alpes, La Tronche, Isere
  - Centre Francois Baclesse, Caen, Normandy
  - Centre Hospitalier Universitaire De Poitiers, Poitiers, Nouvelle-Aquitaine
  - Nantes University Hospital, Nantes, Pays de la Loire Region
  - Hopital Ambroise Pare, Boulogne
  - CHU Estaing, Clermont-Ferrand
  - Regional University Hospital of Lille 2208, Lille
  - Hopital Timone, Marseille
  - Centre Hospitalier Universitaire De Nice Hopital De L Archet, Nice
  - Saint Louis Hospital, Paris, Île-de-France Region
  - Gustave Roussy, Villejuif, Île-de-France Region
- Germany (17):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - LMU Klinikum, Munich, Bavaria
  - University Hospital of Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - University Hospital Giessen, Giessen, Hesse
  - Elbekliniken Stade Buxtehude, Buxtehude, Lower Saxony
  - Muhlenkreiskliniken Minden, Ruhr University Bochum, Bochum, North Rhine-Westphalia
  - University Hospital Essen, Essen, North Rhine-Westphalia
  - Hautklinik, Ludwigshafen am Rhein, Rhineland-Palatinate
  - University Hospital Dresden, Dresden, Saxony
  - Universitatsklinikum Leipzig, AoR, Leipzig, Saxony
  - Universitatsklinikum Schleswig Holstein Campus Luebeck, Lübeck, Schleswig-Holstein
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - SRH Wald- Klinikum Gera GmbH, Gera, Thuringia
  - Charite University Medicine, Berlin
  - Klinikum Bremen Ost, Bremen
- Italy (11):
  - Azienda Ospedaliera Santa Croce i Carle, Cuneo
  - Azienda Ospedaliero-Universitaria Ferrara, Ferrara
  - Fondazione IRCCS Istituto Nazionale dei Tumori., Milan
  - Istituto Europeo di Oncologia, Milan
  - Universita della Campania Luigi Vanvitelli, Naples
  - Istituto Nazionale Tumori IRCCS Fondazione G Pascale, Napoli
  - Azienda Ospedaliero-Universitaria Maggiore della Carita - Oncology, Novara
  - U.O. Oncologia Medica 2 Universitaria, Azienda Ospedaliero Universitaria Pisana, Pisa
  - Campus Bio-Medico di Roma, Rome
  - Medical Oncology, Taormina
  - Azienda Sanitaria Universitaria del Friuli Centrale, Udine
- Spain (13):
  - Hospital Universitario Virgen de las Nieves, Granada, Andalusia
  - Hospital Universitario Virgen De La Victoria Malaga, Málaga, Andalusia
  - Hospital Universitari Son Espases, Palma, Balearic Islands
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Instituto Oncologico Dr Rosell, Barcelona, Catalonia
  - Hospital Clinico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Vall d'Hebron Hospital, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Clinico Universitario San Cecilio, Granada
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Instituto Valenciano de Oncologia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/